CLINICAL TRIAL: NCT06045520
Title: Effects of Information-Motivation-Behavioral Skills Model on Disease Management of Adolescents With Epilepsy: Randomized Controlled Study
Brief Title: Effects of Information-Motivation-Behavioral Skills Model on Disease Management of Adolescents With Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Ozlem Guzel Polat, PhD (c), Nursing, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MersinU-HB-OGP-02
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Nursing Caries
Keywords: adolescent; epilepsy; education training; pediatric nursing; Information-Motivation-Behavioral Skills Model
MeSH Terms: conditions — Epilepsy | interventions — Information Motivation Behavioral Skills Model

STUDY DESIGN:
Intervention Model Description: The research has a randomized controlled interventional study design. An impartial investigator who is not participating in the study will conduct the randomization. Six alternative combinations with a block size of four (ABAB(1), ABBA(2),...) containing codes A and B will be constructed using the block randomization method. From 1 to 6, combinations will be numbered. By sorting the integers (1-6) via randomizer.org 33 times in a random order, a random assignment sequence will be formed. By drawing lots with coins, it will be established which of the A and B codes is the intervention group and which is the control group. Participants who meet the inclusion criteria will be asked to sign an informed consent form, and their group will be shared with the researcher after the pre-tests (T1) are completed. In the intervention group, participants will get a web-based training based on the family-centered approach.
Who Masked: Participant
Masking Description: The participants were unaware of which group they were assigned to. The data will be entered using A and B codes, and the researcher doing the statistical analysis will be blind to the participants' groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBM Educational Training (Experimental): Intervention group participants will receive IBM skills model on educational training intervention for 8 weeks.
  Interventions: Behavioral: Information-Motivation-Behavioral Skills Model
- Control Group (No Intervention): No intervention was applied to the control group.

INTERVENTIONS:
Behavioral: Information-Motivation-Behavioral Skills Model — 1.-2.Meeting:Regarding the information component of the IMB model; Answers given by the adolescents to the epilepsy knowledge test, the topics on which the adolescent wants to get information will be agreed with the adolescent and an education training will be created.3.,4.,5.-6. Meeting:Personal motivation, which is the first step of the motivation component; A meeting will be held regarding the obstacles to the disease, attitudes and behaviors towards the disease. In order to strengthen social support systems, a one-session seizure management training will be planned with a person chosen by the adolescent from his parent or friend group.7-8. Meeting:Seizure self-efficacy and treatment compliance will be evaluated in the behavioral skills component. During training, achievable goals will be set to ask the adolescent to provide personal feedback, ask open-ended questions, engage in reflective listening, and increase personal and social motivation to comply with medical recommendations
  Arms: IBM Educational Training

SUMMARY:
The adolescent's search for self-discovery and identity in physical, psychosocial, cognitive and emotional areas may become more complex with epilepsy disease management. The adolescent's burden of treatment compliance may lead to poor adherence to the disease and worsen short- and long-term health outcomes. Disease self-management in epilepsy represents the processes required for disease knowledge, seizure control, medication adherence, increasing social support and quality of life, and reducing the negative effects of the disease. Educational training implemented in this period have an effect that increases motivation to gain skills to adapt to the disease. This model argues that knowledge is a basis for behaviour change, but it is not sufficient alone. However, it is argued that people will have the necessary behavioural skills when they are well informed and motivated for effective action. It is aimed to find a statistically significant difference from the scales (Epilepsy Knowledge Test for Adolescents, Seizure Self-Efficacy Status Scale in Children with Epilepsy, Multidimensional Perceived Level of Social Support Scale, Child's Attitude Towards His/her Disease Scale) at the end of the training of adolescents who received an 8-week training program.

DETAILED DESCRIPTION:
Research Hypotheses H1: There is a difference between the seizure self-efficacy scale scores of the intervention group based on the IMB model and the control group.

H2: There is a difference between perceived social support of scale scores of the intervention group based on the IMB model and the control group.

H3: There is a difference between child attitude towards illness scale scores of the intervention group based on the IMB model and the control group.

H4: There is a difference between knowledge test for epilepsy disease scale scores of the intervention group based on the IMB model and the control group.

Epilepsy is the most common neurological disease in childhood. Due to the diagnosis in childhood, parents take a more active role in disease management, while the child remains more passive in this process. In this period, the burden of adaptation of the parents to the treatment passes to the adolescent who is in the process of transition from childhood to adulthood. The adolescent's search for self-discovery and identity in physical, psychosocial, cognitive and emotional areas may become more complex with epilepsy disease management. The adolescent's burden of treatment compliance may lead to poor adherence to the disease and worsen short- and long-term health outcomes. Disease self-management in epilepsy represents the processes required for disease knowledge, seizure control, medication adherence, increasing social support and quality of life, and reducing the negative effects of the disease. Adolescents have low personal motivation for disease management and therefore need more social support from parents and peers. Educational training implemented in this period have an effect that increases motivation to gain skills to adapt to the disease. Fisher et al. developed the IBM model in order to develop health behaviour for HIV prevention in adolescents. This model argues that knowledge is a basis for behaviour change, but it is not sufficient alone. However, it is argued that people will have the necessary behavioural skills when they are well informed and motivated for effective action. In the studies conducted, it was determined that the fact that the model was simple, understandable, low cost and clearly defined implementation stages supported adolescents to develop health behaviour skills. When the international and national literature was examined, no training based on the Knowledge Motivation Behaviour model for adolescents with epilepsy was found. The fact that the model is simple, understandable, low cost and clearly defined implementation stages will support the disease management of adolescents. It is thought that adolescents who are well informed and well motivated with the training based on the Knowledge Motivation Behaviour model and who have developed behavioural skills with training can support disease management.

IMPLEMENTATION OF RESEARCH

Data will be collected in the pediatric neurology department of a university hospital in the Mediterranean region of southern Turkey. Patients and their parents who meet the inclusion criteria will be informed about the study and the education training. Verbal consent will be obtained by the researcher from the patient who agrees to participate in the study. Pre-test forms (Epilepsy Knowledge Test for Adolescents, Seizure Self-Efficacy Status Scale in Children with Epilepsy, Multidimensional Perceived Level of Social Support Scale, Child's Attitude Towards His/her Disease Scale) will be applied. After the forms are administered, the assignment sequence, registration of the participants and patients will be assigned to the intervention or control groups by an independent researcher.

Written informed consent will then be obtained from patients assigned to the intervention and control groups and their parents. Adolescents with epilepsy in the intervention group will receive an 8-session educational training. Each session will be limited to 10-12 adolescents and the intervention group will be divided into three groups of 11. Each session of the training will be limited to 40-50 minutes. The researchers are working as a lecturer in the departments of pediatric health and diseases nursing and pediatric neurology and as a specialist nurse with a total of 14 years of experience in the neonatal intensive care unit and paediatric health and diseases service. Sessions will be held with the participation of at least one of the researchers.

Sessions will be held with the participation of at least one researcher. The training program was developed by researchers and program development specialists. Within the scope of the research, a separate session on seizure management will be held for an individual requested by the adolescents in order to increase the social support level of the adolescents. Post-test forms (Epilepsy Knowledge Test for Adolescents, Seizure Self-Efficacy Status Scale in Children with Epilepsy, Multidimensional Perceived Social Support Level Scale, Child's Own Illness Scale) were administered to the adolescents in the intervention group immediately after completing the 8-session training program and one month later (twice in total). Towards Attitude Scale) will be applied again.

Informed written consent forms will be obtained from the adolescents in the control group and their parents immediately after they accept the research, and pre-test forms (Epilepsy Knowledge Test for Adolescents, Seizure Self-Efficacy Status Scale in Children with Epilepsy, Multidimensional Perceived Social Support Level Scale, Child's Attitude Towards His Own Illness Scale. ) will be applied. After the pre-test forms are applied, no intervention will be applied to the control group. .

Adolescents in the control group will not receive any intervention other than standard care and routine monitoring provided by the doctor and nurse at the outpatient clinic. Immediately after the training program given to the adolescents in the intervention group was completed and one month later (twice in total), post-test forms were administered to the control group (Epilepsy Knowledge Test for Adolescents, Seizure Self-Efficacy Status Scale in Children with Epilepsy, Multidimensional Perceived Social Support Level Scale, Child's Self-Efficacy Scale). Attitude Towards Illness Scale) will be administered again.

After the data collection phase, after the analysis of the data and determining that the training program is effective, the training program will be applied to the control group without any changes in the training program given to the intervention group.

STATISTICAL

A statistical package program will be used in the analysis of the data. The conformity of the mean scores of the scale to the normal distribution will be evaluated with the coefficients of kurtosis and skewness, and the means will be compared with parametric or nonparametric test techniques. The similarity of the groups in terms of demographic and clinical characteristics will be evaluated with the relevant tests. Cohen's d effect size will be calculated to express the size of the difference between the means.

ELIGIBILITY:
Inclusion Criteria:

For adolescents;

* Those who agree to participate in the study and sign the Informed Voluntary Consent Form
* Age between 12-18 years
* Diagnosis of epilepsy
* No communication barriers (visual, hearing, mental retardation)
* No other chronic disease other than epilepsy
* Being literacy

Exclusion Criteria:

For adolescents;

* Refusal to participate in the study
* Those who do not sign the Informed Volunteer Consent Form
* Those who do not sign the Informed Volunteer Consent Form
* Under 12 years old, over 18 years old,
* No diagnosis of epilepsy
* Communication disability (visual, hearing, mental retardation)
* No another chronic disease other than epilepsy
* Illiteracy

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-06-08 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Change in the mean score of adolescents in the epilepsy disease knowledge test | an average of 3 month
  The "epilepsy knowledge test for adolescents" developed by the researchers consists of 25 items. The knowledge test includes true and false items. The items were evaluated with item prop. correct and item discrimination index ITEMAN analysis. The reliability coefficient, which provides evidence of the internal consistency of the knowledge test, was found to be KR-20 (Kuder-Richardson) = 0.813.
Change in the mean score of adolescents in the Seizure Self-Efficacy Scale in Children with Epilepsy | an average of 3 month
  The scale, which was developed by Caplin et al. and whose Turkish validity and reliability study was conducted by Güven and İşler in 2015, is a 15-item 5-point Likert-type scale. It was conducted with children aged 9-18 years with epilepsy and the cronbach alpha value was found to be 0.89. The scale is a 15-item five-point Likert-type scale and the scale items are scored between 1-5. A high score on the scale is interpreted as an improved seizure self-efficacy of the child
Change in the mean score of adolescents in the Multidimensional Perceived Social Support Scale | an average of 3 month
  The Multidimensional Perceived Social Support Scale was developed by Zimet et al. The Cronbach's alpha coefficient of the scale, whose validity and reliability study was performed by Eker et al. in 2001, was found to be 0.80-0.95. The scale consists of 12 items and evaluates social support received from three different sources. The scale consists of a 7-point Likert scale as "Absolutely no 1,2,3,4,5,5,6,7 Absolutely yes". The scale has a total of three sub-dimensions as family (mother, father, spouse, children and siblings), friend and special person support (dating, oral, fiancé, neighbour, relative, doctor) and each sub-dimension consists of 4 items. The sub-dimension scores are obtained by summing the four items in the sub-dimensions, and the total score is obtained by summing all sub-dimensions. A minimum score of 12 points and a maximum score of 84 points can be obtained from the scale. A high total score indicates a high level of perceived social support
Change in the mean score of adolescents in theChild's Attitude Towards His Own Illness Scale | an average of 3 month
  The Turkish validity and reliability study of the scale developed by Austin and Huberty was conducted by Ersun and Bolışık. The scale, whose Cronbach Alpha value is 0.79, is a 5-point Likert type and consists of 15 items. The original scale was developed for children aged 8-12 with chronic diseases. However, in a systematic review of the scale, it was stated that it could be used safely between the ages of 8 and 22. 4 of the 13 items are bipolar adjectives (Very Good, Somewhat Good, Not Sure, Somewhat Bad, Very Bad) and 9 are from options expressing how often they experience the positive and negative aspects of having a chronic disease (Very Often, Often, Sometimes , Not Often, Never). Among the scale items scored between 1 and 5, 1 and 2 indicate negative attitude, 3 indicate neutral attitude, and 4 and 5 indicate positive attitude.

CONTACTS AND LOCATIONS:
Overall Officials: Ayda Çelebioğlu, Study Director — Mersin University
Locations (1):
- Mersin University, Mersin, Turkey (Türkiye)

REFERENCES:
- [Background] Tutar Guven S, Isler Dalgic A, Duman O. Evaluation of the efficiency of the web-based epilepsy education program (WEEP) for youth with epilepsy and parents: A randomized controlled trial. Epilepsy Behav. 2020 Oct;111:107142. doi: 10.1016/j.yebeh.2020.107142. Epub 2020 Jul 21. PMID 32702651
- [Background] Fisher JD, Amico KR, Fisher WA, Harman JJ. The information-motivation-behavioral skills model of antiretroviral adherence and its applications. Curr HIV/AIDS Rep. 2008 Nov;5(4):193-203. doi: 10.1007/s11904-008-0028-y. PMID 18838059
- [Background] Fisher JD, Fisher WA, Williams SS, Malloy TE. Empirical tests of an information-motivation-behavioral skills model of AIDS-preventive behavior with gay men and heterosexual university students. Health Psychol. 1994 May;13(3):238-50. doi: 10.1037//0278-6133.13.3.238. PMID 8055859
- [Background] Lerch MF, Thrane SE. Adolescents with chronic illness and the transition to self-management: A systematic review. J Adolesc. 2019 Apr;72:152-161. doi: 10.1016/j.adolescence.2019.02.010. Epub 2019 Mar 21. PMID 30903932
- [Background] Braga P, Mifsud J, D'Souza C, Clarke M, Honein A, Tovuudorj A, Pfafflin M. Education and epilepsy: Examples of good practice and cooperation. Report of the IBE Commission on Education. Epilepsy Behav. 2020 Feb;103(Pt A):106653. doi: 10.1016/j.yebeh.2019.106653. Epub 2019 Nov 21. PMID 31761687